CLINICAL TRIAL: NCT05221528
Title: Study on the Association Between Lipid Profiles and Cardiovascular Events: Analysis From the Korean Nationwide Health Insurance Database
Brief Title: Association Between Lipid Profiles and Cardiovascular Events
Acronym: KORLIPID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Mo Yang, MD, PhD, Seoul National University Hospital
Other Study IDs: E-2101-012-1184
Record Dates: First submitted 2021-10-28; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemias; Cardiovascular Diseases
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of lipid profiles — Measured: total cholesterol, high-density lipoprotein cholesterol, and triglyceride Calculated: low-density lipoprotein

SUMMARY:
KORLIPID (Study on the Association between Lipid Profiles and Cardiovascular Events) registry enrolled 4234339 subjects who underwent general health check-ups provided by National Health Insurance Service in 2009.

DETAILED DESCRIPTION:
Subjects who underwent general health check-ups provided by National Health Insurance Service in 2009 were included in KORLIPID study. Demographic data, anthropometric data and medical information from general health check-ups were collected. In addition, medical records in National Health Insurance Service between 2002 and 2018 were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent general health check-ups in 2009

Exclusion Criteria:

* Age less than 30 years
* Age 75 years or more

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects (age 30-74 years) who underwent general health check-ups in 2009
Sampling Method: Probability Sample
Enrollment: 4234339 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2023-01-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarction | until 2018 after inclusion
  acute myocardial infarction demanding hospitalization

SECONDARY OUTCOMES:
Stroke | until 2018 after inclusion
  acute ischemic stroke demanding hospitalization
Heart failure | until 2018 after inclusion
  acute heart failure demanding hospitalization
Death | until 2018 after inclusion
  all cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
For reasonable request, data are available through approval and oversight by the Korean national health insurance service.